CLINICAL TRIAL: NCT03469414
Title: Manual Wheelchair Speed, Maneuverability, and Endurance and Community Access
Status: Terminated | Type: Observational
Why Stopped: COVID-19 Pandemic made participant recruitment nonfeasible.
Sponsor: Allina Health System (Other)
Responsible Party: Sponsor
Other Study IDs: CKNF-1703
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Physical Disability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Wheelchair Mobility and Speed: This group will participate in activity-based measures employed in routine occupational and physical therapy practice to assess participants' wheelchair speed, maneuverability, and endurance. These measures include: the Life Space Assessment Scale, 6-Minute Push Test, Forward Push Test, Wheelchair Slalom Test, Craig Handicap Assessment and Reporting Technique, and PART-O.
  Interventions: Other: Life Space Assessment Scale; Other: 6-Minute Push Test; Other: Forward Push Test; Other: Wheelchair Slalom Test; Other: Craig Handicap Assessment and Reporting Technique; Other: PART-O
- GPS Tracking: A GPS tracker will be placed on the wheelchairs of 25 individuals who consent to participate in this arm of the project. Using a GPS tracker will provide a direct measure of the community locations these participants go. The GPS location is collected every minute, and mapped to Google Maps, which would allow calculation of speed of movement.
  Interventions: Other: Life Space Assessment Scale; Other: 6-Minute Push Test; Other: Forward Push Test; Other: Wheelchair Slalom Test; Other: Craig Handicap Assessment and Reporting Technique; Other: PART-O; Other: GPS Tracking

INTERVENTIONS:
Other: Life Space Assessment Scale — This nine question survey asks participants where they have gone in the last week, frequency of those visits, and how independently they went there.
Other: 6-Minute Push Test — The 6 Minute Push Test is a measure of endurance, and requires that the participant wheel themselves around two pylons that are located 15 meters apart for 6 minutes.
Other: Forward Push Test — This measure of wheelchair propulsion speed asks patients to propel themselves as fast as they can over 20 meters. This task is performed twice, and the average time is used for the score.
Other: Wheelchair Slalom Test — In this measure, participants propel themselves through an 18 meter slalom course at their maximum self-selected speed, wheeling around seven cones, separated by three, two, or one meter.
Other: Craig Handicap Assessment and Reporting Technique — A measure of social participation in individuals with SCI.
Other: PART-O — The PART-O is a community participation measure.
Other: GPS Tracking — A GPS tracker will be attached to the wheelchairs of a subset of participants for one week. The GPS location is collected every minute, and mapped to Google Maps, which would allow calculation of speed of movement.
  Groups: GPS Tracking

SUMMARY:
This is a cross-section correlational study that will examine the relationships between wheelchair speed, maneuverability, and endurance with community integration. By identifying which of these has the biggest contribution to community participation, the information will be used to justify continues therapy, to alter the focus of therapy, and to justify purchase of power or power assist wheelchairs when needed. Currently, therapists make the recommendation for a power or power assist chair based on their clinical judgement and the patient's experience, but there has been limited justification from the literature for these decisions. Finally, because the CHART measure is the gold standard in rehabilitation research for community integration, but has psychometric problems, we will use this opportunity to validate a new more psychometrically solid measure, the PART-O, against the CHART.

ELIGIBILITY:
Inclusion criteria include:

* 18 years or older
* presence of a physical disability
* use of a manual wheelchair for primary mobility
* living in the community.

Exclusion criteria would include:

* individuals who have significant expressive or receptive language deficits (i.e. aphasia, verbal apraxia, etc.)
* limb orthopedic conditions that would contraindicate speed and endurance testing, such as recent fractures or joint instability
* cardiopulmonary resting heart rate of less than 50 or over 100, resting vitals of systolic blood pressure of > 200 or < 90, diastolic blood pressure of >110, resting O2 levels of less than 90 (ACSM, 205; Fletcher, et al., 1993).
* any other cardiac symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 260 participants with disabilities who use manual wheelchairs for their primary mobility. Participants will be recruited from all Courage Kenny Rehabilitation Institute sites. Participants will have a mixture of diagnosis, with a minimum of 30 individuals with diagnosis of stroke and 30 individuals with diagnosis with spinal cord injury.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-03-31 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Life Space Assessment Scale Score | Day 0
  This nine question survey asks participants where they have gone in the last week, frequency of those visits, and how independently they went there. The locations vary from spaces within their home, immediately around their home, or outside of their neighborhood, city, county, state or nation. Their independent movement patterns will be classified as within the home, limited community mobility and full community mobility.

SECONDARY OUTCOMES:
Distance (meters) covered in six-minute push test | Day 0
  This is a measure of endurance, and requires that the participant wheel themselves around two pylons that are located 15 meters apart for 6 minutes
Average time to complete forward push test | Day 0
  This measure of wheelchair propulsion speed asks patients to propel themselves as fast as they can over 20 meters. This task is performed twice, and the average time is used for the score
Time to complete Manual Wheelchair slalom Test | Day 0
  In this measure, participants propel themselves through an 18 meter slalom course at their maximum self-selected speed, wheeling around seven cones, separated by three, two, or one meter

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Flinn, PhD, OTR/L, Principal Investigator — Allina Health
Locations (1):
- Courage Kenny Rehabilitation Institute, Golden Valley, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No